CLINICAL TRIAL: NCT02510105
Title: Tomodensitometric Study of Pulmonary Effects of Intrapulmonary Percussive Ventilation in ARDS Patients
Acronym: PERVE-ARDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0236
Record Dates: First submitted 2015-06-01; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: ARDS
Keywords: Critical Care; ARDS; Intrapulmonary Percussive Ventilation; VDR4; Lung aeration; CT scan
MeSH Terms: interventions — Tomography, X-Ray Computed; Intubation

ARMS (1):
- ARDS patients (Experimental)
  Interventions: Device: VDR4 ventilator (Intrapulmonary Percussive Ventilation); Device: CT scan; Device: Servo-i; Device: - Intubation; Device: Ventilation ( with an ICU conventional ventilator)

INTERVENTIONS:
Device: VDR4 ventilator (Intrapulmonary Percussive Ventilation)
Device: CT scan
Device: Servo-i
Device: - Intubation
Device: Ventilation ( with an ICU conventional ventilator)

SUMMARY:
The study is intended to elucidate the pulmonary effects of Intrapulmonary Percussive Ventilation (IPV) with VDR4 ventilator of patients with ARDS, using computed tomography (CT).

DETAILED DESCRIPTION:
Prospective clinical study in ICU of ventilated patients with ARDS. The morphologic pulmonary effects of IPV with VDR4 are not known to the investigators' knowledge.

The main aim is to quantify recruited, normally aerated and overinflated parts of the lungs after a 1 hour treatment with IPV.

Patients with ARDS (focal and non focal) consecutively admitted to the investigators' ICU are enrolled after informed consent.

Patients are intubated and ventilated with Servo-I (GE) and ventilation is optimized according to ARDS-network recommandations.

A first thoracic CT-scan is performed with ICU ventilator and then the patient is ventilated with VDR4 during 1 hour.

A second thoracic CT-scan is then performed and the patient re-ventilated with ICU ventilator.

Arterial blood gases and hemodynamic parameters are recorded during experiments.

CT-scan are analysed and compared for normally aerated, overinflated and recruited lung parenchyma. Regions are determined thanks to their Hounsfield units (HU).

ELIGIBILITY:
Inclusion Criteria:

* Patients ventilated more than 48 h
* Sedated patients
* ARDS moderate or severe (Berlin 2012)
* Patients who have given their consent or his family
* Patients aged between 18 and 85 years

Exclusion Criteria:

* Pregnant ou lactating women
* Hemodynamic instability
* Chronic respiratory insufficiency.
* Pneumothorax
* Fistulae bronchopleural

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (H0) in volume of overinflated lung at H1 | at Hour 0(just before Intrapulmonary Percussive Ventilation) and Hour 1(just after Intrapulmonary Percussive Ventilation)

SECONDARY OUTCOMES:
Volume of normally aerated lung | at Hour 0 (just before Intrapulmonary Percussive Ventilation ) and Hour 1 (just after Intrapulmonary Percussive Ventilation)
Volume of recruited lung | at day 1 (between H0 and H1)
Heart rate | at day 1 ((every 10 min between H0 and H1)
Blood pressure | at day 1 (every 10 min between H0 and H1)
Arterial blood gaz | at day 1 ((every 10 min between H0 and H1)
Evolution of catecholamine doses (µg/Kg/min) | at day 1 (every 10 min between H0 and H1)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel CONSTANTIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Godet T, Jabaudon M, Blondonnet R, Tremblay A, Audard J, Rieu B, Pereira B, Garcier JM, Futier E, Constantin JM. High frequency percussive ventilation increases alveolar recruitment in early acute respiratory distress syndrome: an experimental, physiological and CT scan study. Crit Care. 2018 Jan 11;22(1):3. doi: 10.1186/s13054-017-1924-6. PMID 29325586